CLINICAL TRIAL: NCT05879224
Title: Feasibility of High Daily Dose Short Course Primaquine After G6PD Testing for the Radical Cure of Plasmodium Vivax Malaria
Brief Title: Short Course Primaquine for the Radical Cure of P. Vivax Malaria - Indonesia
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Gadjah Mada University (Other); Universitas Sumatera Utara (Other); Indonesia University (Other); Yayasan Pengembangan Kesehatan dan Masyarakat (Unknown); Indonesian National Malaria Control Program, Ministry of Health (Unknown); National Research and Innovation Agency of Indonesia (Unknown); Burnet Institute (Other); University of Melbourne (Other); Medicines for Malaria Venture (Other); PATH (Other); UNITAID (Other); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MMV_PQ_21_01 U1111-1291-3218
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Vivax Malaria; G6PD Deficiency
Keywords: Primaquine
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Intervention Model Description: Combination Product: Revised case management package
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Revised case management package (Experimental)
  Interventions: Combination Product: Revised case management package

INTERVENTIONS:
Combination Product: Revised case management package — 1. Point-of-care quantitative G6PD testing using G6PDSTANDARD (SD Biosensor) prior to use of primaquine (Day 0)
  2. Prescription of short course primaquine (7 mg/kg total)(Day 0):
     * PQ7 (1 mg/kg/day for 7 days) if G6PD activity greater than 70 percent
     * PQ14 (0.5 mg/kg/day for 14 days) if G6PDactivity is 30-70 percent
     * PQ8w (0.75 mg/kg/week for 8 weeks) if G6DPactivity less than 30 percent
  3. Participant counselling at the health facility (Day 0):
     * Supervision of first dose of primaquine
     * Education regarding the importance and risks of primaquine therapy and necessity to take primaquine with food
  4. Community based clinical review on Day 3 (and Day 7 for the first 300 participants) to detect and manage gastrointestinal or haemolytic adverse effects of treatment and encourage adherence to full treatment regime
  5. Improved malariometric surveillance and pharmacovigilance to support wider scale use of the revised case management

SUMMARY:
The proportion of malaria that is the Plasmodium vivax species is increasing in Indonesia. Reducing vivax malaria will require innovative solutions to cure both the blood and liver stages of the disease. This study will evaluate of the feasibility of implementing point-of-care glucose-6-phosphate dehydrogenase deficiency (G6PD) testing. This will be followed by high dose, short course primaquine treatment regimens for patients with vivax malaria, and combined with patient education, surveillance, and pharmacovigilance. We plan to implement the study at 6 health facilities across Indonesia using a staged before-and-after study, with a mixed method evaluation.

DETAILED DESCRIPTION:
Significant gains have been made in reducing the overall burden of malaria worldwide, however these have been far greater for Plasmodium falciparum than P. vivax. P. vivax remains a major obstacle to malaria control and elimination efforts, largely due to its ability to form dormant liver stages (hypnozoites) that allow it to escape detection and treatment. Importantly, they are susceptible only to 8 aminoquinolines such as primaquine however, primaquine is associated with risk of haemolysis in individuals with a genetic condition, called glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Additionally, the recommended 14-day prolonged treatment regimen is associated with poor treatment adherence hence ineffective primaquine treatment. Innovative solutions to the radical cure of both the blood and liver stages of P. vivax are urgently required.

The Indonesian Ministry of Health has requested a pragmatic study of the feasibility and cost-effectiveness of implementing point-of-care G6PD testing followed by high-dose, short-course primaquine treatment regimens for patients with vivax malaria. These interventions are to be combined with practicable enhancements to patient education, supervision, malariometric surveillance and pharmacovigilance.

This will be a before-after longitudinal health facility-based study implemented at six sites in Indonesia; four in Papua, one in North Sumatra and one in Lampung. We will use a staged approach for the implementation of the revised case management strategy, including patient education and counselling,community-based clinical review, with mixed methods evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vivax malaria

Exclusion Criteria:

* Patients who are pregnant
* Patients who are breastfeeding
* Patients with a Hb <8g/dL
* Patients with a previous adverse reaction to primaquine
* Patient with severe malaria

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2999 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing at least one Serious Adverse Event (SAE) during treatment | During treatment (up to 8 weeks) ]
  SAEs are collected during clinical review using a study-specific questionnaire
Proportion of patients experiencing at least one Adverse Event of Special Interest(AESI) during treatment | During treatment (up to 8 weeks)
  AESIs (haemolysis, methaemoglobinaemia and gastrointestinal discomfort) are collected during clinical review using a study-specific questionnaire
Proportion of patients with P. vivax malaria who correctly receive all components of the revised case management package | 3 days
  Measured by completion of G6PD testing and the correct prescription of primaquine based on G6PD activity, completion of patients counselling and community based follow up on Day 3

SECONDARY OUTCOMES:
The proportion of patients with any AESI during treatment | During treatment (up to 8 weeks)
  AESIs are collected during clinical review using a study-specific questionnaire
The proportion of patients with a gastrointestinal (GI) AESI during treatment | During treatment (up to 8 weeks)
  AESIs are collected during clinical review using a study-specific questionnaire
The proportion of patients with an AESI related to haemolysis during treatment | During treatment (up to 8 weeks) ]
  AESIs are collected during clinical review using a study-specific questionnaire
The proportion of patients an AESI related to methaemoglobinaemia | During treatment (up to 8 weeks)
  AESIs are collected during clinical review using a study-specific questionnaire
Proportion of patients permanently stopping PQ before end of treatment | During treatment (up to 8 weeks)
  Discontinuation of PQ will be assessed using a study-specific questionnaire
The proportion of patients receiving correct treatment based on G6PD activity | 1 day
  This will be assessed by linking patients G6PD activity results measured during study enrolment with primaquine dose prescribed on the same day
Proportion of patients who were reviewed on Day 3 and Day 7 | 1 week
  This will be assessed by linking patients enrolment data with Day 3 and Day 7clinical review data
Perception of and experience with new radical cure tools among health care providers and community members | 6 months
  This will be assessed using stakeholder interviews
Proportion of health care practitioners who comply with the revised radical cure treatment algorithm | 1 day
  The outcome will be assessed from patients' enrolment data
Proportion of patients receiving a SD Biosensor G6PD test | 1 day
  The outcome will be assessed from patients' enrolment data
Proportion of eligible P. vivax malaria patients receiving the correct dose of primaquine based on the result of the G6PD test | 1 day
  The outcome will be assessed from patients' enrolment data
Proportion of P. vivax malaria patients who are ineligible for daily primaquine and are incorrectly given primaquine (including infants, pregnant females and G6PD deficient patients | 1 day
  The outcome will be assessed from patients' enrolment data
Proportion of P. vivax malaria patients that are reviewed on Day 3 | 3 days
  This will be assessed by linking patients' enrolment data with clinical review data
Proportion of P. vivax malaria patients that adhere to their prescribed primaquine regimen | 3 days
  This will be assessed by linking patients' enrolment data with clinical review data
Factors influencing acceptability and feasibility of the new radical cure tools among health care providers are identified | 3 days
  This will be assessed using stakeholder interviews, observations and focus groups
Barriers and enablers of uptake and implementation at the sub-national levels are identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Factors influencing compliance with G6PD testing and perceptions of new drug regimens and serious adverse events among health care providers are identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Required knowledge, skills, and training to administer the revised case management and patient-counselling identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Factors influencing the barriers and facilitators to patient adherence to primaquine after the rollout of the revised case management identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Factors influencing the acceptability and feasibility of community-based clinical review at Day 3 of primaquine treatment identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Perceptions of the new radical cure tools and serious adverse events at the community level identified | 18 months
  This will be assessed using stakeholder interviews and focus groups
Local acceptability of the revised case management algorithms among patients, their families, and healthcare workers established | Day 3
  This will be assessed using stakeholder interviews and focus groups
The monthly incidence of confirmed symptomatic P. vivax malaria episodes (mono-infection or mixed) before implementation versus after implementation | 18 months
  This will be assessed by comparing facility surveillance data before implementation with facility surveillance data after implementation
The prevalence of P. vivax parasitaemia in patients presenting with fever before implementation versus after implementation | 18 months
  This will be assessed by comparing cross-sectional data on n=200 patients (per facility) collected before implementation to the prevalence collected in n=200patients (per facility) after implementation
Cumulative risk of representation to the same clinic with symptomatic P. vivax malaria within 6 months | 18 months
  This will be assessed by linking patients' enrolment data
Costs of implementing policy from a healthcare provider perspective, including health systems strengthening processes | 18 months
  This will be assessed from health system data collected throughout the study
Household costs per P. vivax episode | 3 days
  This will be assessed from a household cost survey on a subset of patients
Overall cost-effectiveness of changing policy if revised case management is effective | 18 months
  This will be assessed from health system data collected throughout the study
Cost per episode of P. vivax malaria from the healthcare provider and societal perspectives | 18 months
  This will be assessed from health system data collected throughout the study
Cost per component of the revised case management package | 18 months
  This will be assessed from health system data collected throughout the study
If revised case management package is effective (significantly reduces the incidence of malaria), then the cost-effectiveness of implementing the revised case management as compared with usual care | 18 months
  This will be assessed from health system data collected throughout the study
Proportion of CHWs who correctly act on early signs of haemolytic anaemia and GI events (i.e. refer patients for further medical review, instruct patient to discontinue treatment) | 3 days
  This will be assessed from clinical review data and study-specific questionnaire
Number of patients with an SAE who are identified by community or clinic staff follow-up and referred to hospital for further management | During treatment (up to 8 weeks)
  This will be assessed by linking clinical review data, study specific questionnaire and SAE form
The proportion of patients eligible to receive PQ who had a SAE during treatment | During treatment (up to 8 weeks)
  This will be assessed by linking enrolment data, clinical review, study specific questionnaire and SAE form
Prevalence of severe anaemia in patients presenting with fever before and after implementation | 18 months
  This will be assessed by comparing the facility surveillance data before implementation with facility surveillance data after implementation

CONTACTS AND LOCATIONS:
Overall Officials: Ric Price, MD, Principal Investigator — Menzies School of Health Research
Locations (6):
- Indonesia (6):
  - Puskesmas Hanura, Hanura, Lampung
  - Puskesmas Tanjung Leidong, Labuhanbatu, North Sumatra
  - Puskesmas Bhintuka, Mimika, Special Region of Papua
  - Puskesmas Pasar Sentral, Mimika, Special Region of Papua
  - Puskesmas Timika, Mimika, Special Region of Papua
  - Puskesmas Wania, Mimika, Special Region of Papua

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be made available to others. The results will be published in peer-reviewed open access journals and disseminated to stakeholders. De-identified quantitative data for the purposes of confirming risk of adverse events will be available to researchers who provide a methodological sound proposal that is in line with the aims of the approved protocol.
Supporting Information: Study Protocol, SAP
Access Criteria: Access is subject to approval by the SCOPE Data Access Committee to ensure that the use of data protects the interests of the participants and researchers according to the terms of ethics approval and principles of equitable data sharing. Requests can be submitted to the Requests can be submitted to Professor Ric Price, Menzies School of Health Research, Email:ric.price@menzies.edu.au and Dr Jeanne Rini Poespoprodjo, Universitas Gadjah Mada, Email:didot2266@yahoo.com

REFERENCES:
- [Derived] SCOPE Study Group. High daily dose Short COurse PrimaquinE after G6PD testing for the radical cure of Plasmodium vivax malaria in Indonesia and Papua New Guinea: the SCOPE implementation study protocol. BMC Infect Dis. 2025 Jul 16;25(1):922. doi: 10.1186/s12879-025-11109-9. PMID 40670924